CLINICAL TRIAL: NCT05799898
Title: Fast-Track Cardiovascular Assessment for Suspicion of Cardiovascular Events on Immunecheckpoint Inhibitors: Prospective Cohort Study.
Brief Title: Fast-Track Cardiovascular Assessment for Suspicion of Cardiovascular Events on Immunecheckpoint Inhibitors
Acronym: FAST-TRACK
Status: Recruiting | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIO-03-2022
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Immune Checkpoint Inhibitor; Cardiovascular Complication; Immune-related Adverse Event
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endomyocardial biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention for research purposes only — No intervention for research purposes only

SUMMARY:
Prospective study cohort on patients addressed for suspected cardiovascular event on immune checkpoint inchibitors.

Longitudinal prospective single center cohort. Inclusion criteria: all patient willing to particiupate seen in the cardio-oncology unit at our institution for the suspicion of heart failure, atherosclerosis related event, Tako Tsubo, arrhymias, pericarditis, myocarditis on antiPD1, antiPDL1, or antiCTLA4 immune checkpoint inhibitors.

Description of patients characteristics, investigations, diagnosis after multidisciplinary meeting, outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all patient referred to the cardio oncology unit for suspected immune related cardiovascular complication on immune checkpoint inhibitors

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults on immune checkpoint inhibitors for cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular event | 12 months
  Composite endpoint: acute coronary syndrome, myocarditis, pericarditis, heart failure, Taki Tsubo, ventricvular arrhymias

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Mirabel, MD, PhD, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Intitut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided